CLINICAL TRIAL: NCT01660854
Title: Re-exposure of Previously Immunized and Challenged Human Volunteers to a Heterologous Strain of P. Falciparum Sporozoites
Brief Title: Re-exposure of Human Volunteers to a Heterologous Strain of P. Falciparum Sporozoites
Acronym: TIP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TIP4
Record Dates: First submitted 2012-07-23; First posted 2012-08-09 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2012-07

CONDITIONS: Malaria, Falciparum
Keywords: Plasmodium; falciparum; malaria; heterologous; immunity
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Proguanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heterologous challenge (Experimental): Biological: Heterologous challenge with 5 infected mosquito bites (NF135) after previous CPS immunization and challenge.
  Drug: Malarone treatment When thick smear positive, of at day 21 after challenge, all volunteers will be treated with malarone.
  Other Name: atovaquone/proguanil
  Interventions: Biological: Heterologous challenge; Drug: Malarone treatment
- Challenge control (Active Comparator): Biological: Plasmodium falciparum mosquito challenge by the bites of 5 Plasmodium falciparum infected mosquitoes (NF135).
  Drug: Malarone treatment When thick smear positive, of at day 21 after challenge, all volunteers will be treated with malarone.
  Other Name: atovaquone/proguanil
  Interventions: Biological: Heterologous challenge; Drug: Malarone treatment

INTERVENTIONS:
Biological: Heterologous challenge — challenge by the bites of 5 Plasmodium falciparum infected mosquitoes.
Drug: Malarone treatment — Three days: 4 tablets 250/100mg per day
  Other Names: atovaquon/proguanil

SUMMARY:
In a previous study (NL33904.091.10) the investigators challenged 24 volunteers after Chloroquine Prophylaxis Sporozoites (CPS) immunization with 45, 30 or 15 infected mosquito-bites respectively. The availability of this immunized cohort opens the unique opportunity to determine protection to a heterologous challenge for both of the protected and unprotected volunteers as the previous challenge infection might have served as immunological boost to the unprotected volunteers.

In the current observational, proof of principle study, the investigators aim to investigate the protection on an individual basis of these previously immunized and challenged volunteers against a heterologous P. falciparum challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 35 years healthy volunteers (males or females)
2. Good health based on history and clinical examination
3. Negative pregnancy test
4. Use of adequate contraception for females
5. Signing of the informed consent form, thereby demonstrating understanding of the meaning and procedures of the study
6. Agreement to inform the general practitioner and to sign a request to release medical information concerning contra-indications for participation in the study
7. Willingness to undergo a Pf controlled challenge through mosquito bites
8. Agreement to stay in a hotel room close to the trial centre during a part of the study (Day 5 after challenge till treatment is finished)
9. Reachable (24/7) by mobile phone during the whole study period
10. Available to attend all study visit
11. Agreement to refrain from blood donation to Sanquin or for other purposes, during the whole study period
12. Willingness to undergo HIV, hepatitis B and hepatitis C tests
13. Negative urine toxicology screening test at screening visit and the day before challenge
14. Willingness to take a curative regimen of Malarone®

Exclusion Criteria:

1. History of malaria (other than participation in ZonMw1 study) or residence in malaria endemic areas within the past six months
2. Plans to travel to malaria endemic areas during the study period
3. Plans to travel outside of the Netherlands during the challenge period
4. Previous participation in any malaria vaccine study and/or positive serology for Pf (except ZonMw1 volunteers)
5. Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
6. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
7. History of arrhythmias or prolonged QT-interval
8. Positive family history in 1st and 2nd degree relatives for cardiac events < 50 years old
9. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
10. Clinically significant abnormalities in electrocardiogram (ECG) at screening
11. Body Mass Index (BMI) below 18 or above 30 kg/m2
12. Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
13. Positive HIV, HBV or HCV tests
14. Participation in any other clinical study within 30 days prior to the onset of the study
15. Enrollment in any other clinical study during the study period
16. For women: being pregnant or lactating
17. Volunteers unable to give written informed consent
18. Volunteers unable to be closely followed for social, geographic or psychological reasons
19. History of drug or alcohol abuse interfering with normal social function
20. A history of treatment for psychiatric disease
21. A history of convulsions
22. Contra-indications to Malarone®, including hypersensitivity or treatment taken by the volunteer that interferes with Malarone®
23. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids and oral anti-histaminic are allowed) and during the study period
24. Any confirmed or suspected immunosuppressive or immunodeficient condition, including (functional) asplenia
25. Co-workers or trainees of the departments Infectious Diseases, Medical Microbiology or Parasitology of the Leiden University Medical Centre (LUMC) or Medical Microbiology, Parasitology, Radboud University Nijmegen (RUNMC)
26. A history of sickle cell anaemia, sickle cell trait, thalassaemia (or trait), G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Duration of prepatent period after challenge infection as measured by microscopy | 21 days after challenge

SECONDARY OUTCOMES:
• Parasitemia and kinetics of parasitemia as measured by PCR | 21 days after challenge
Frequency of signs or symptoms in study groups | 21 days after challenge
• Immune responses between study groups | 21 days after challenge

CONTACTS AND LOCATIONS:
Overall Officials: RW Sauerwein, PhD, Study Director — Radboud University Medical Center
Locations (1):
- Leiden University Medical Centre, Leiden, Leiden, Netherlands

REFERENCES:
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Derived] Schats R, Bijker EM, van Gemert GJ, Graumans W, van de Vegte-Bolmer M, van Lieshout L, Haks MC, Hermsen CC, Scholzen A, Visser LG, Sauerwein RW. Heterologous Protection against Malaria after Immunization with Plasmodium falciparum Sporozoites. PLoS One. 2015 May 1;10(5):e0124243. doi: 10.1371/journal.pone.0124243. eCollection 2015. PMID 25933168